CLINICAL TRIAL: NCT01929044
Title: A Randomized, Double-blind, Independent 3rd Party Unblind, Active-controlled, Parallel-group, Multi-center Trial, in Contrast With Anisodamine (654-II), 10mg, to Evaluate the Efficacy and Safety of Buscopan® Solution for Injection, 20mg (Intramuscularly) for the Treatment of Acute Gastric or Intestinal Spasm-like Pain
Brief Title: Efficacy of Buscopan® in Comparison With 654-II (Anisodamine) in Acute Gastric or Intestinal Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202.848
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-01

CONDITIONS: Intestinal Diseases
MeSH Terms: conditions — Intestinal Diseases | interventions — anisodamine; Butylscopolammonium Bromide

ARMS (2):
- Buscopan® (hyoscine butylbromide) (Experimental): 1st injection of Buscopan® solution 20mg, if necessary 2nd injection after 20min of the 1st injection
  Interventions: Drug: Buscopan® (hyoscine butylbromide)
- 654-II(anisodamine) (Active Comparator): 1st injection of 654-II solution 10mg, if necessary 2nd injection after 20min of the 1st injection
  Interventions: Drug: 654-II (anisodamine)

INTERVENTIONS:
Drug: 654-II (anisodamine) — 10mg injection
  Arms: 654-II(anisodamine)
Drug: Buscopan® (hyoscine butylbromide) — 20mg injection
  Arms: Buscopan® (hyoscine butylbromide)

SUMMARY:
The aim of the study is to assess the efficacy of Buscopan® (hyoscine butylbromide) in comparison to 654-II (anisodamine)in acute gastric or intestinal spasm-like pain.

ELIGIBILITY:
Inclusion criteria:

1. Patients must sign and date an Informed Consent consistent with International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines and local regulation prior to participation in the trial.
2. Patients must agree to cooperate with all trial evaluations and perform all required tasks.
3. Patients with acute gastric or intestinal spasm-like pain (without severe vomiting and surgical acute abdomen).
4. Male or female patients aged 18 to 70 years.
5. The pain intensity upon screening is at least point 6 on a 0-10 numerical rating scale (NRS).

Exclusion criteria:

1. Patients with the following concomitant disease is not eligible for enrollment:

   * Painful gastric or intestinal spasm of organic origin such as Crohn's disease, ulcerative colitis, lactose intolerance, gastrointestinal perforation, suspected gastrointestinal perforation or peritoneal effusion.
   * Pain related with malignancy.
   * Patients with other severe pain states of organic origin.
   * Mechanical stenosis of the gastrointestinal tract ,megacolin.
   * Urinary retention associated with mechanical stenosis of urinary tract.
   * Narrow-angled glaucoma.
   * Tachyarrhythmia.
   * Myasthenia gravis.
   * Meulengracht-Gilbert syndrome.
   * Known depression or known mental illness, anxiety disturbance.
2. Patients taking the following concomitant medication within 7 half-life of concomitant medication (the duration from taking concomitant medication to attending the trial is less than 7 half-life) are not eligible for enrollment:

   * Analgesics,
   * Spasmolytics,
   * Anticholinergics
   * Affecting gastrointestinal motility, such as propantheline, metoclopramide, cisapride, loperamide, diphenoxylate, opioid analgesics, antacids and other ulcer treatment
   * Regular administration of laxatives
   * Narcotics
   * Antidepressant treatment or treatment with psychoactive drugs
3. Pregnancy and/or lactation or planned pregnancy;
4. Known hypersensitivity to N-butylscopolammonium bromide
5. Alcohol, or drug abuse.
6. Simultaneous participating in another clinical trial, or discontinuing from another clinical trial before randomization (administration of study medication); moreover, in the case of screening failure or premature discontinuing from the trial, repeated enrollment is forbidden.
7. Unwilling to or unable to complete the entire trial procedure according to the protocol.
8. In investigator's opinion, the patient is not proper for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- China (20):
  - 202.848.86016 Boehringer Ingelheim Investigational Site, Baotou
  - 202.848.86008 Boehringer Ingelheim Investigational Site, Beijing
  - 202.848.86009 Boehringer Ingelheim Investigational Site, Beijing
  - 202.848.86010 Boehringer Ingelheim Investigational Site, Beijing
  - 202.848.86013 Boehringer Ingelheim Investigational Site, Beijing
  - 202.848.86012 Boehringer Ingelheim Investigational Site, Changchun
  - 202.848.86020 Boehringer Ingelheim Investigational Site, Changsha
  - 202.848.86018 Boehringer Ingelheim Investigational Site, Chenzhou
  - 202.848.86007 Boehringer Ingelheim Investigational Site, Chongqing
  - 202.848.86021 Boehringer Ingelheim Investigational Site, Chongqing
  - 202.848.86006 Boehringer Ingelheim Investigational Site, Guangzhou
  - 202.848.86003 Boehringer Ingelheim Investigational Site, Hangzhou
  - 202.848.86022 Boehringer Ingelheim Investigational Site, Huanggang
  - 202.848.86001 Boehringer Ingelheim Investigational Site, Shanghai
  - 202.848.86011 Boehringer Ingelheim Investigational Site, Shanghai
  - 202.848.86015 Boehringer Ingelheim Investigational Site, Shenyang
  - 202.848.86014 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 202.848.86019 Boehringer Ingelheim Investigational Site, Wenzhou
  - 202.848.86004 Boehringer Ingelheim Investigational Site, Wuhan
  - 202.848.86005 Boehringer Ingelheim Investigational Site, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 299 patients were entered and 295 were treated.
Groups:
- Buscopan® (Hyoscine Butylbromide): Single intramuscular injection of 20 mg Buscopan® solution (if needed, second injection with 20 mg was to be made at 20 min after the first one) was administered to the patients
- 654-II (Anisodamine): Single intramuscular injection of 10 mg Anisodamine solution (if needed, second injection with 10 mg was to be made at 20 min after the first one) was administered to the patients
Period: Overall Study
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Started | 153 | 146
Completed | 142 | 129
Not Completed | 11 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 9 | 14
Not completed — Not Treated | 1 | 3

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomised patients who received at least one dose of study medication constituted the treated set. One patient was randomized to 654-II but incorrectly treated with Buscopan® so in the disposition table and efficacy analysis, number of patients are 152 and 143 while for demographic and AE analysis, they are 153 and 142.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine) | Total
Number analyzed (Participants) | 153 | 142 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (14.2) | 40.7 (14.8) | 41.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 76 | 166
  Male | 63 | 66 | 129

OUTCOME MEASURES:

1. Primary Outcome: PID From Pre-dose Baseline at 20 Minutes After First Injection.
Description: Pain intensity difference (PID) from pre-dose baseline at 20 minutes after first injection. It was assessed using an 11-point numerical rating scale (NRS) ranging from 0 = 'no pain' to 10 = 'worst pain possible'.
Time Frame: Baseline and 20 minutes after the first injection
Population: Per-Protocol Set (PPS): All patients in full analysis set (FAS: all patients who provided any data for the primary efficacy endpoint constituted the full analysis set.), who revealed no important protocol violations that would impact the analysis of primary endpoint
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Units on a scale | -4.09 (0.17) | -3.66 (0.18)
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Restricted maximum likelihood (REML) -repeated measures approach; Test type: Non-Inferiority or Equivalence — One-sided test relative to the non-inferiority margin of 1; p < 0.0001, Mixed Models Analysis; Kenward-Roger approximation is used to estimate the denominator degrees of freedom. An unstructured covariance matrix is used; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.88 to 0.04], Standard Error of Mean 0.23 — REML-based repeated measures approach includes baseline pain intensity as continuous covariate, treatment, centre, time and treatment-time interaction as fixed effects. The difference was calculated as Buscopan minus 654-II
Statistical Analysis 2: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0743, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.88 to 0.04], Standard Error of Mean 0.23 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: PID From Pre-dose Baseline at 10 Minutes After First Injection.
Description: Pain intensity difference (PID) from pre-dose baseline at 10 minutes after first injection. It was assessed using an 11-point numerical rating scale (NRS) ranging from 0 = 'no pain' to 10 = 'worst pain possible'.
Time Frame: Baseline and 10 minutes after the first injection
Population: Per-Protocol Set (PPS): All patients in full analysis set (FAS), who revealed no important protocol violations that would impact the analysis of primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Units on a scale | -2.64 (0.14) | -2.33 (0.15)
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.1210, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.70 to 0.08], Standard Error of Mean 0.20 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: PID From Pre-dose Baseline at 30 Minutes After First Injection.
Description: Pain intensity difference (PID) from pre-dose baseline at 30 minutes after first injection. It was assessed using an 11-point numerical rating scale (NRS) ranging from 0 = 'no pain' to 10 = 'worst pain possible'.
Time Frame: Baseline and 30 minutes after the first injection
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Units on a scale | -5.14 (0.15) | -4.74 (0.16)
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0658, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.82 to 0.03], Standard Error of Mean 0.21 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: PID From Pre-dose Baseline at 60 Minutes After First Injection.
Description: Pain intensity difference (PID) from pre-dose baseline at 60 minutes after first injection. It was assessed using an 11-point numerical rating scale (NRS) ranging from 0 = 'no pain' to 10 = 'worst pain possible'.
Time Frame: Baseline and 60 minutes after the first injection
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Units on a scale | -5.96 (0.14) | -5.51 (0.15)
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0220, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.85 to -0.07], Standard Error of Mean 0.20 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: PID From Pre-dose Baseline at 120 Minutes After First Injection.
Description: Pain intensity difference (PID) from pre-dose baseline at 120 minutes after first injection. It was assessed using an 11-point numerical rating scale (NRS) ranging from 0 = 'no pain' to 10 = 'worst pain possible'.
Time Frame: Baseline and 120 minutes after the first injection
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Units on a scale | -6.46 (0.13) | -6.01 (0.14)
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.81 to -0.09], Standard Error of Mean 0.18 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Global Assessment of Efficacy by the Patient at 120 Minutes After the First Injection
Description: Global assessment of efficacy by the patient. The patient was to assess the efficacy at 120 min after the first injection using a 4-point rating scale by answering the question: "How would you rate the effect of the study medication for relieving your acute gastric or intestinal spasm-like pain?" (0 = poor; 1 = fair; 2 = good; 3 = very good).
Time Frame: 120 minutes after the first injection
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Percentage of Patients
  Very Good | 22.5 | 22.0
  Good | 59.2 | 44.1
  Fair | 18.3 | 29.1
  Poor | 0.0 | 4.7
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0113, van Elteren test; The van Elteren test stratifying for centre (Cochran-Mantel-Haenszel test using modified ridit scores) was performed

7. Secondary Outcome: Proportion of Patients Who Need the Second Injection
Description: Proportion of patients who need the second injection at 20 minutes after the first injection.
Time Frame: 20 minutes after the first injection.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Number analyzed (Participants) | 142 | 127
Percentage of Patients | 24.6 [17.81 to 32.58] | 33.9 [25.70 to 42.79]
Statistical Analysis 1: Comparison: Buscopan® (Hyoscine Butylbromide) vs 654-II (Anisodamine); Test type: Superiority or Other; p = 0.0992, Regression, Logistic; A logistic regression model was used to evaluate the response with treatment as fixed effect and baseline pain intensity as continuous covariate; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.37 to 1.09] — Exact 95% confidence interval obtained by Clopper and Pearson approach

ADVERSE EVENTS:
Time Frame: From first study drug application until 2 days (inclusive) after the last study drug application
Arm/Group | Buscopan® (Hyoscine Butylbromide) | 654-II (Anisodamine)
Serious Adverse Events (participants affected / at risk) | 1/153 | 0/142
Other Adverse Events (participants affected / at risk) | 12/153 | 10/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buscopan® (Hyoscine Butylbromide) (N=153) | 654-II (Anisodamine) (N=142)
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buscopan® (Hyoscine Butylbromide) (N=153) | 654-II (Anisodamine) (N=142)
Thirst (General disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.